CLINICAL TRIAL: NCT00139282
Title: A Phase 3, Multicenter, Randomized, Double-Masked, Controlled Study of Squalamine Lactate (MSI-1256F) for Injection for the Treatment of Subfoveal Choroidal Neovascularization Associated With Age-Related Macular Degeneration
Brief Title: A Safety and Efficacy Study of Squalamine Lactate for Injection (MSI-1256F) for "Wet" Age-Related Macular Degeneration
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Genaera Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSI-1256F-301
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2007-11-28 (Estimated); Status verified 2007-11

CONDITIONS: "Wet" Age-Related Macular Degeneration
Keywords: wet AMD; macular degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — squalamine lactate

INTERVENTIONS:
Drug: Squalamine Lactate

SUMMARY:
Age-Related Macular Degeneration (AMD) is a degenerative eye disease of the retina that causes a progressive loss of central vision. AMD is the leading cause of blindness among adults age 50 or older in the Western world. AMD presents in two different types: "dry" and the more severe "wet" form. Wet AMD is caused by the growth of abnormal blood vessels in the macula. Squalamine lactate is an investigational drug that may prevent the growth of these abnormal blood vessels. This study will evaluate the safety and efficacy of Squalamine lactate in the treatment of AMD in patients, the exact number of which will be determined based on data from the sponsor's ongoing Phase 2 trials.

The trial objective is to evaluate the safety and efficacy of two doses of Squalamine lactate for Injection administered as intravenous infusions weekly for 4 weeks followed by maintenance doses every 4 weeks through week 104 compared with the safety and efficacy in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of "wet" age-related macular degeneration

Exclusion Criteria:

* Prior treatment for "wet" age-related macular degeneration in the affected eye in the past 3 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-06

PRIMARY OUTCOMES:
Loss in best corrected visual acuity (BCVA) of greater than or equal to 15 letters (ETDRS) at 52 weeks in the study eye compared to baseline.

SECONDARY OUTCOMES:
Change in retinal thickness in the study eye at 52 and 104 weeks compared to baseline, as measured by OCT, in a subset of subjects
Change in area of CNV in the study eye at 52 and 104 weeks compared to baseline, as measured by fluorescein angiography
Gain or loss in BCVA of greater than or equal to 15 letters (ETDRS) at 52 and 104 weeks in the fellow eye compared to baseline in the subgroup of subjects whose fellow eye is affected with wet AMD
Loss in binocular visual acuity of greater than or equal to 15 letters at 52 and 104 weeks compared to baseline, using a modified ETDRS protocol.

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Eldorado Retina Associates, Louisville, Colorado
  - Florida Eye Microsurgical Institute, Boynton Beach, Florida
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - University of Florida, Jacksonville, Florida
  - Magruder Eye Institute, Orlando, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Retina Associates of Florida, Tampa, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Midwest Eye Institute, Indianapolis, Indiana
  - Retina Associates, PA, Shawnee Mission, Kansas
  - Cumberland Valley Retina Consultants, PC, Hagerstown, Maryland
  - Delaware Valley Retina Associates, Lawrenceville, New Jersey
  - Retina Associates of New Jersey, Teaneck, New Jersey
  - MaculaCare, New York, New York
  - Charlotte Eye, Ear, Nose & Throat Associates, Charlotte, North Carolina
  - Horizon Eye Care, Charlotte, North Carolina
  - The Ohio State University, Havener Eye Institute, Columbus, Ohio
  - Penn State Ophthalmology, Hershey, Pennsylvania
  - Retina Vitreous Consultants, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Genaera Corporation, Plymouth Meeting, Pennsylvania
  - Carolina Retina Center, Columbia, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Southeastern Retina Associates, Kingsport, Tennessee
  - Retina Research Center, Austin, Texas
  - Garcia & Associates, MD, PA, Houston, Texas
  - John Moran Eye Center, Salt Lake City, Utah
  - Virginia Retina Center, Leesburg, Virginia